CLINICAL TRIAL: NCT01540435
Title: Perioperative FOLFOXIRI and Bevacizumab Compared With Postoperative FOLFOX in Patients With Resectable Liver Metastases From Colorectal Cancer (PERIMAX). A Randomized, Multidisciplinary DGAV(CAO-V/CALGP)/AIO Phase II Trial
Brief Title: Perioperative Treatment of Resectable Liver Metastases
Acronym: PERIMAX
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University of Regensburg (Other)
Collaborators: University of Halle Medical Faculty (Other)
Responsible Party: Principal Investigator, Hans J Schlitt, Prof. MD, Principal Investigator, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KKSH088; 2010-023575-25 (EudraCT Number)
Record Dates: First submitted 2012-02-16; First posted 2012-02-28 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Colon Cancer Liver Metastasis
Keywords: Colorectal cancer; Liver metastases; Perioperative treatment; Liver resection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postoperative Arm (Arm A) (No Intervention): FOLFOX:
  Oxaliplatin at a dose of 85 mg/m2 iv over two hours (day 1) I-LV at a dose of 200 mg/m2 iv over two hours (day 1) 5-FU at a dose of 3200 mg/m2 iv over 48 hours (day 1-3)
  Duration of treatment:
  Treatment will be administered for 12 cycles (6 months) postoperatively starting 6 weeks after surgery.
- Perioperative Arm (Arm B) (Experimental): Therapy will be administered in a biweekly schedule. First preoperative cycle will be administered with 75% of dosage for FOLFOXIRI, if no diarrhea ≥ grade 3 occurs, following cycles should be administered in full dosage.
  FOLFOXIRI + bevacizumab:
  bevacizumab at a dose of 5 mg/kg iv over 30 to 90 min (day 1) irinotecan at a dose of 165 mg/m2 iv over two hours (day 1) oxaliplatin at a dose of 85 mg/m2 iv over two hours (day 1) I-LV at a dose of 200 mg/m2 iv over two hours (day 1) 5-FU at a dose of 3200 mg/m2 iv over 48 hours (day 1-3)
  Duration of treatment:
  Treatment will be administered for 6 cycles (3 months) preoperatively (last cycle without bevacizumab), after 6 weeks followed by liver surgery, after further 6 weeks followed by 6 cycles (3 months) postoperatively.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab at a dose of 5 mg/kg iv over 30 to 90 min (day 1) + FOLFOXIRI in a biweekly schedule, 6 cycles preoperatively, 6 cycles postoperatively
  Other Names: VEGF antibody
  Arms: Perioperative Arm (Arm B)

SUMMARY:
This randomized, controlled, multicenter, non-comparative phase II trial compares an intensified perioperative treatment of patients with resectable synchronous or metachronous colorectal liver metastases to primary surgery and adjuvant systemic chemotherapy.

DETAILED DESCRIPTION:
Recurrence rates after R0-resection of colorectal liver metastases are still very high (about 60-70 %). Therefore, multidisciplinary treatment of these patients is frequently used in order to achieve a beneficial impact regarding progression-free and overall survival. The point in time of treatment, pre- and/or postoperative, is still a matter of debate. In the EORTC 40983 trial, perioperative chemotherapy with 5-Fluorouracil and oxaliplatin (FOLFOX-Regimen) displayed a non-significant benefit in 3 year disease free survival in the intent to treat population (HR 0.79, 95% CI 0.62 to 1.02) (Nordlinger, Sorbye et al. 2008). The combined analysis of two adjuvant trials, with a (non-contemporary) 5-FU Bolus regimen, showed a non-significant prolongation of median disease free survival (DFS) from 18.8 to 27.9 months (p=0.058) and OS from 47.3 to 62.2 months (p=0.095) (Mitry, Fields et al. 2008). However, postoperative treatment with 6 months of FOLFOX is often used in daily practise. Thus, further investigation is urgently warranted.

This phase II trial evaluates two strategies with intensified perioperative or postoperative treatment regimens. Current studies established the role of the FOLFOXIRI regimen in the metastatic setting (Falcone, Ricci et al. 2007). A further intensification of a three drug regimen with bevacizumab seem to be feasible yielding response rates up to 84% and a disease control rate up to 100% (Falcone 2008; Bruera, Santomaggio et al. 2010; Masi, Loupakis et al. 2010). Regarding the efficacy, evaluation of FOLFOXIRI and bevacizumab in preoperative treatment for resectable CLM seems to be promising. Postoperative treatment with FOLFOX for 6 months was chosen for arm A.

ELIGIBILITY:
Main selection criteria:

1. Histological proven CRC with completely resectable metachronous or synchronous liver metastases (as judged by the treating surgeon).
2. Patients must have undergone complete resection (R0) of the primary tumor at least 4 weeks before randomization. Or in case of synchronous disease with intact primary; the primary tumor have to be R0 resectable together with the liver metastases and the patient has a non-obstructive primary tumor and is able to receive preoperative chemotherapy before surgery. Synchronous rectal primary is not allowed.
3. Measurable hepatic disease by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
4. No evidence of extra-hepatic metastasis of CRC.
5. Patients must be from 18 to 75 years.
6. ECOG Performance status ≤ 1
7. No previous chemotherapy for metastatic disease. Radiotherapy alone is allowed if given pre or post protocol treatment.
8. Previous adjuvant chemotherapy for primary CRC is allowed if completed at least 6 months before inclusion in this study.
9. All the following tests should be done within 4 weeks prior to randomization

   * Absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L, and hemoglobin > 9 g/dL or 5.59 mmol/l.
   * Serum creatinine less than 1.5 times the upper limit of normal (ULN) (to exclude severe renal impairment); no significant proteinuria (urine dipstick for proteinuria ³ 2+. If urine dipstick is ³ 2+, 24-hour urine must demonstrate £ 1 g of protein in 24 hours for patient to be eligible).
   * Absence of major hepatic insufficiency (bilirubin < 1.5 x ULN and aspartate aminotransferase (ASAT)/alanine aminotransferase (ALAT) < 5 x ULN).
   * Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and aPTT < 1.5 ULN within 7 days prior to registration. The use of full dose anticoagulants is allowed as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least two weeks at the time of registration.
10. No pregnancy or breast feeding. Negative serum pregnancy test within 7 days of starting study treatment in pre-menopausal women and women < 1 year after the onset of menopause is required before entering in the trial. Note: a negative test has to be reconfirmed by a urine test, should the 7-day window be exceeded.
11. Adequate contraception is required during and for 3 months after study treatment for both male and female patients if the risk of conception exists.
12. No major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to randomization.
13. No previous exposure to VEGF/VEGFR-targeting therapy within the last 12 months.
14. No thrombosis or severe bleeding within 6 months prior to entry into the study (except for bleeding of the tumor before its surgical resection) and no evidence of bleeding diathesis or coagulopathy.
15. Absence of peripheral neuropathy NCI CTCAE-grade ≥ 1, active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as > 4 loose stools per day), serious wound complications, ulcers, or bone fractures.
16. No evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
17. No concomitant treatment with ASS > 325 mg or NSAIDs, known to inhibit platelet function, sorivudin or analog compounds or preparations of St. John's wort.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Failure-free survival (FFS@18) | 18 months
  Failure will be defined as no R0 resection, local or distant recurrence or death from any cause.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 5 years
Overall survival (OS) | 5 years
Perioperative morbidity | 30 days (hospital stay)
Quality of life | 12 months
Achievability of R0 resection | intraoperative
Overall response rate (Arm B) | 3 months
Pathologic response rate | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans J. Schlitt, Prof. MD, Study Chair — Department of Surgery, University Medical Center Regensburg; Hans-Joachim Schmoll, Prof. MD, Study Director — Department of Internal Medicine IV, University Hospital Halle

REFERENCES:
- [Background] Stein A, Glockzin G, Wienke A, Arnold D, Edelmann T, Hildebrandt B, Hollerbach S, Illerhaus G, Konigsrainer A, Richter M, Schlitt HJ, Schmoll HJ. Treatment with bevacizumab and FOLFOXIRI in patients with advanced colorectal cancer: presentation of two novel trials (CHARTA and PERIMAX) and review of the literature. BMC Cancer. 2012 Aug 16;12:356. doi: 10.1186/1471-2407-12-356. PMID 22897915